CLINICAL TRIAL: NCT06206707
Title: Faecal Microbiota Transplantation for Immune Checkpoint Inhibitor-mediated Diarrhea/Colitis: a Randomised, Double-blind Pilot Efficacy and Safety Study
Brief Title: FMT in Checkpoint Inhibitor-mediated Diarrhea and Colitis
Acronym: Immunobiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-10-72-105-23
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Diarrhea; Colitis; Malignant Melanoma; Kidney Cancer
MeSH Terms: conditions — Diarrhea; Colitis; Melanoma; Kidney Neoplasms | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo controlled, randomised trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faecal microbiota transplantation (FMT) (Experimental): Patients receive two applications of capsule FMT with 3-7 days between applications.
  Interventions: Procedure: Faecal Microbiota Transplantation (FMT)
- Placebo (Placebo Comparator): Patients receive two applications of placebo capsules with 3-7 days between applications.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Faecal Microbiota Transplantation (FMT) — Capsule FMT
  Other Names: Fecal Microbiota Transplantation; FMT
  Arms: Faecal microbiota transplantation (FMT)
Procedure: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the outcome of patients with immune checkpoint inhibitor-mediated diarrhea/colitis (IMC) treated with faecal microbiota transplantation (FMT) in a randomised, placebo-controlled trial.

The aim of the present study is to assess the feasibility, pilot efficacy, and safety of FMT for patients with IMC.

Participants will be treated two times with capsule FMT or placebo capsules in a 1:1 ratio. The intervention treatment will be an add-on to the patients' standard treatment for IMC.

Researchers will compare the FMT-treated group to the placebo-treated group to see if FMT promotes remission of IMC.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above.
2. Histologically proven diagnosis of malignant melanoma and/or kidney cancer.
3. Treatment with any immune checkpoint inhibitor (Nivolumab, Pembrolizumab, Cemiplimab, Atezolizumab, Durvalumab, Avelumab, Ipilimumab), alone or in combination, within the last 8 weeks.
4. Grade 2 or higher CTCAE diarrhea, of which at least 3 stools are Bristol chart score 6-7.
5. Negative PCR for enteric pathogens including C. difficile, after the onset of diarrhea.
6. Signed written informed consent.

Exclusion Criteria:

1. Diagnosed bacterial infection requiring antibiotic treatment at inclusion.
2. Pregnancy or breastfeeding. Pregnancy ruled out by male sex, postmenopausal women or a negative choriogonadotropin (hCG) urine test.
3. Primary diarrheal disease pre-existing to the immune checkpoint inhibitor treatment, including inflammatory bowel disease.
4. Unable to ingest capsules.
5. Unable to understand written or oral patient information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission of immune-mediated diarrhea | At 42 days after intervention treatment
  Number of patients with steroid-free resolution of diarrhea, defined as < 3 liquid stools (Bristol <6) per 24 hours during day 40 and 41 after the last intervention treatment.

SECONDARY OUTCOMES:
Remission of diarrhea defined by CTCAE | At 42 days after intervention treatment
  Number of patients in steroid-free clinical remission of diarrhea 6 weeks (42 days) after the last intervention treatment. Clinical remission is defined as < 4 stools over baseline per day (CTCAE diarrhea grade 1 or less), at day 40 and 41.
Remission of colitis defined by CTCAE | At 42 days after intervention treatment
  Number of patients in steroid-free clinical remission of colitis 6 weeks (42 days) after the last intervention treatment. Clinical remission is defined as asymptomatic in regards to colitis (CTCAE colitis grade 1 or less), at day 40 and 41.
Therapy response of FMT | Up to 12 weeks after intervention treatment
  Therapy response defined as a decrease of at least 3 points in Simple Clinical Colitis Activity Index (SCCAI) score, at weeks 1, 6 and 12 after the last intervention treatment.
Number of days until CTCAE diarrhea grade 1 | Up to 12 weeks after intervention treatment
  Number of days until less than 4 stools over baseline per day (CTCAE diarrhea grade 1 or less), lasting a minimum of 48 consecutive hours with no increase in steroid dose in the 12 weeks of follow-up.
Number of days until resolution of diarrhea | Up to 12 weeks after intervention treatment
  Number of days until resolution of diarrhea, defined as 3 or fewer Bristol type 6-7 stools per day, lasting a minimum of 48 consecutive hours.
Incidence of fecal microbiota transplantation (FMT)-related adverse events | At 42 days after intervention treatment
  Number of adverse events (AE) during first 6 weeks after intervention treatment. AE's will be graded by CTCAE.
Incidence of fecal microbiota transplantation (FMT)-related serious adverse events | At 12 weeks after intervention treatment
  Number of serious adverse events (SAE) during 12 weeks follow-up after the final intervention treatment. SAE's will be graded by CTCAE.
Faecal microbiota composition | Up to 6 weeks after intervention treatment
  Changes in faecal microbiome composition from baseline to week 6 after the last intervention.
Gut mucosa-associated microbiome | Up to 6 weeks after intervention treatment
  Changes in mucosa-associated microbiome from baseline to week 6 after the last intervention.
Faecal-calprotectin | Up to 6 weeks after intervention treatment
  Percentual change in faecal-calprotectin from prior to intervention to week 6 after the last intervention.
Blood immunological parameters | Up to 6 weeks after intervention treatment
  Changes in blood immunological parameters (including circulating cytokines) from baseline and at week 6 after the last intervention.
Hospitalisation | Up to 12 weeks after intervention treatment
  Hospitalisation defined as the total number of days hospitalised, during 12 weeks of follow-up.
Colectomy | Up to 12 weeks after intervention treatment
  Colectomy during 12 weeks of follow-up.
Mortality | Up to 12 weeks after intervention treatment
  Mortality during the 12 weeks of follow-up.
Accumulated steroid dose | Up to 12 weeks after intervention treatment
  Accumulated steroid dose (total dose in mg) during 12 weeks following experimental treatment.
Resumption of immune checkpoint inhibitor therapy | Up to 12 weeks after intervention treatment
  Number of patients resuming immune checkpoint inhibitor therapy during the 12 weeks of follow-up.
Response to immune checkpoint inhibitor therapy | Up to 12 weeks after intervention treatment
  Response to immune checkpoint inhibitor therapy defined by Response Evaluation Criteria in Solid Tumours (RECIST 1.1 and iRECIST).
Patient and physician perceptions of FMT treatment | At 42 days after intervention treatment
  Patient and physician perceptions of FMT treatment and the usage for IMC assessed by a patient questionnaire at week 6 and a physician questionnaire.
Health-related quality of life | At 42 days after intervention treatment
  Changes in health-related quality of life assessed by EQ-5D-5L at baseline and week 6.
Endoscopic response | Up to 6 weeks after intervention treatment
  Endoscopic response, defined as decrease in Mayo endoscopic score ≥1 grade, at week 6 after the last intervention treatment.
Endoscopic remission | Up to 6 weeks after intervention treatment
  Endoscopic remission, defined as Mayo endoscopic score 0, at week 6 after the last intervention treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Hvas, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Open access publication, raw data available upon reasonable request and according to data protection regulation.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Protocol: On request. Other: after study completion
Access Criteria: Evaluated after email request, trnlau@rm.dk

REFERENCES:
- See also: Centre for faecal microbiota transplantation (CEFTA) — https://cefta.au.dk